CLINICAL TRIAL: NCT05192616
Title: Prospective, Multicenter, Non-randomized, Single-arm Observational Study to Evaluate Safety and Effectiveness of iCover Covered Stent for the Treatment of the Aorto-iliac Occlusive Disease
Brief Title: Safety and Effectiveness Evaluation of iCover Covered Stent for the Treatment of the Aorto-iliac Occlusive Disease
Acronym: iliCo
Status: Active, not recruiting | Type: Observational
Sponsor: iVascular S.L.U. (Industry)
Responsible Party: Sponsor
Other Study IDs: iliCo Study
Record Dates: First submitted 2021-12-14; First posted 2022-01-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Angioplasty; Peripheral Arterial Disease; Iliac Artery Disease; Covered Stent; Aorto-Iliac Atherosclerosis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- iCover covered stent: Percutaneous transluminal angioplasty (PTA)
  Interventions: Device: Covered stent implantation

INTERVENTIONS:
Device: Covered stent implantation — Percutaneous transluminal angioplasty (PTA) with iCover covered stent for the treatment of de novo aorto-iliac occlusive lesions

SUMMARY:
The objective of this prospective, multi-center, non-randomized, single-arm observational study is to evaluate the safety and the efficacy of the iCover covered stent over a 24-month follow-up period for the treatment of de novo iliac occlusive lesions, defined by a significant vessel stenosis ≥70%, in patients with symptomatic arteriopathy of the lower limbs (Rutherford class 2 to 5).

DETAILED DESCRIPTION:
This is a prospective, single-arm, multinational, and multicenter study conducted to evaluate the safety and efficacy of the iCover covered stent for the treatment of de novo iliac occlusive lesions (common and/or external iliac arteries) in patients with symptomatic lower limb arteriopathy. The primary endpoint of the study is primary patency, defined as the absence of restenosis in the target lesion over a 12-month follow-up period in patients who did not undergo a reintervention on the target lesion. Restenosis is defined as a reduction in the luminal diameter of more than 50%, assessed either by duplex ultrasound (considered as a peak systolic velocity index ≥ 2.4 at the target lesion) or by angio-CT (multiplanar reconstruction). Secondary endpoints include: technical and procedural success rate, freedom from all major adverse events, incidence of procedure- or device-related major local complications at the treated lesion, rate of SAEs, major amputation rate at the target limb, primary sustained clinical improvement (improvement in Rutherford classification), primary and secondary patency rates, TLR and TVR rates, and changes in ABI, the Walking Impairment Questionnaire, and the EQ-5D questionnaire from baseline.

ELIGIBILITY:
Inclusion criteria

1. ≥ 18 years of age
2. Rutherford clinical stage 2 to 5
3. Significant (≥70%) stenosis of atheromatous iliac lesions evidenced by duplex scan, MRI CT angiography or arteriography
4. De novo atheromatous lesion of the aortoiliac segment
5. Patient informed about the study and collection of the patient's informed consent agreement Exclusion criteria

Subjects will not be eligible to participate in the study if any of the following conditions are present in the subject:

1. Protected adult patients, guardianship, curatorship, safeguard of justice
2. Woman with possibility of pregnancy
3. Patient with asymptomatic atheromatous lesions
4. Patient with inflow lesion in the infrarenal aorta
5. Patient treated with Covered endovascular reconstruction of aortic bifurcation (CERAB reconstruction)
6. Acute ischemia or acute thrombosis
7. Non-atherosclerotic disease
8. History of coagulopathy
9. Severe comorbidities with life expectancy <2 years
10. Contraindication to taking antiplatelet aggregation therapy (aspirin or clopidogrel). The patient must be able to take an antiplatelet aggregation for at least 3 months after the procedure
11. Patient participating in another clinical study which may interfere with the results
12. Comorbidity or any reason which, according to the investigator, could limit the participation, the patient's adherence with the follow-up or the scientific integrity of the study
13. Lesion near or adjacent to an aneurysm
14. Inability to follow-up during the investigation
15. Patient objection to participate in the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic arteriopathy of the lower limbs (Rutherford class 2 to 5). Patients with de novo atheromatous aorto-iliac lesions.
  According to the incidence of TASC II lesions, approximately 70% of the patients will be classified as TASC II A or B lesions, while the other 30% will be classified as TASC II C or D lesions.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Patency | 12 months after index procedure.
  The primary patency, defined as the absence of restenosis in the target lesion over the 12-month follow-up period in patients who did not undergo a reintervention on the target lesion.

SECONDARY OUTCOMES:
Technical success rate | Day 0.
  Technical success rate, defined as the ability to cross and dilate the lesion and achieve residual angiographic stenosis no greater than 30% after iCover stent graft insertion. Outcomes will be computed as the percentage of lesions treated at the end of the procedure.
Procedural success rate | Day 0.
  Procedural success rate, defined as technical success and no complications during the procedure including general and local complications as defined in the protocol. Outcomes will be computed as the percentage of patients at the end of the procedure.
Freedom from All Major Adverse Event (MAEs) | 1, 6, 12, 24 months after index procedure.
  MAEs are described as All-Cause Mortality post-procedure, Target Lesion Revascularization (TLR) post-procedure and Major Amputation of the Target Limb post-procedure (amputations above the ankle of the target leg).
Incidence of Procedure- or Device- related Major Local Complications | Up to 30 days after index procedure.
  Incidence of Procedure- or Device- related Major Local Complications at the treated lesion or Puncture Site up to 30 days post-procedure. Major Local Complications include: Iliac arterial rupture, retroperitoneal hematoma, thrombosis of the iliac axis on the ipsilateral side, need for surgery to achieve hemostasis, bleeding with loss of more than 2 g/ dL of hemoglobin, false aneurysm at the puncture site, preventing resumption of walking at 24 hours or appearance of ischemia on the ipsilateral side.
Rates of Serious Adverse Events (SAEs) | 1, 6, 12, 24 months after index procedure.
  Rates of SAEs, including both related and unrelated events. SAEs will be categorized as related or unrelated to the procedure/device based on adjudication by an Independent Clinical Events Committee.
Major amputation at target limb rate | 1, 6, 12, 24 months after index procedure.
  Percentage of patients with amputations above the ankle of the target leg will be counted.
Primary sustained clinical improvement | 1, 6, 12, 24 months after index procedure.
  Primary sustained clinical improvement defined as a sustained upward shift of 1 category of the Rutherford classification for patients with claudication, and by wound healing and rest pain resolution for patients in critical limb ischemia, without the need for repeated target lesion revascularization in surviving patients.
Primary patency rates | 6 and 24 months after index procedure.
  Primary patency rates, defined as the lack of restenosis without reintervention of the target lesion. Restenosis is defined as a reduction in the luminal diameter of more than 50%, determined by either, duplex ultrasound examination considered as a peak systolic velocity index ≥ 2.4 at the target lesion, or by angio-CT (multiplanar reconstruction). In case of death, the vessel is considered as patent as long as no restenosis was detected during the last visit before the patient died. Outcomes will be computed as the percentage of lesions (Time frame: 6, 24 months after index procedure).
Secondary patency rates | 6, 12, 24 months after index procedure.
  Secondary patency rates, defined as the patency of the stent following an endovascular or surgical reintervention due to significant in-stent restenosis or occlusion. Outcomes computed as percentage of lesions.
Target lesion revascularization (TLR) rate | 1, 6, 12, 24 months after index procedure.
  Target lesion revascularization (TLR) rate, defined as the need for repeated procedures (endovascular or surgical) due to a problem arising from the lesion initially treated in surviving patients with preserved limbs. Outcomes will be computed as the percentage of lesions.
Target vessel revascularization (TVR) rate | 1, 6, 12, 24 months after index procedure.
  Target vessel revascularization (TVR) rate, defined as the need for repeated procedures (endovascular or surgical) due to a problem arising remote from the vessel initially treated in surviving patients with preserved limbs. Outcomes will be computed as the percentage of lesions.
Change in Ankle-Brachial Index (ABI) from baseline | 1, 6, 12, 24 months post-procedure.
  Change in ABI from baseline.
Change in Walking Impairment Questionnaire from baseline | 1, 6, 12, 24 months post-procedure.
  The Walking Impairment Questionnaire values will be recorded and compared to the baseline values. This questionnaire is a validated tool to assess walking capability in patients with Peripheral Arterial Disease in different situations.
Change in quality of life from baseline | 1, 6, 12, 24 months post-procedure.
  Change in quality of life from baseline, as measured by EQ-5D. The EQ-5D Questionnaire values will be recorded and compared to the baseline values. It is a validated questionnaire to measure the quality of life based on 5 different parameters. Worst possible score in this study would be 0, best possible score would be 1. In addition, the patient indicates her/his current health on an analog scale from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Locations (18):
- Belgium (4):
  - Onze Lieve Vrouw Aalst, Aalst
  - Imelda Bonheiden, Bonheiden
  - Az Sint Blasius Dendermonde, Dendermonde
  - ZOL Genk, Genk
- France (5):
  - Centre Hospitalier Universitaire de Brest, Brest
  - CHU Pitié Salpêtrière, Paris
  - Hôpital Paris Saint Joseph, Paris
  - Hôpital privé Saint-Martin, Pessac
  - Hôpital privé Villeneuve d'Ascq, Villeneuve-d'Ascq
- Germany (5):
  - Herzzentrum Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - MVZ Kaiserslautern, Kaiserslautern, Rhineland-Palatinate
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - KEH Berlin, Berlin
  - Imland Klinik Rendsburg, Rendsburg
- Spain (4):
  - Hospital de Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital de Cruces, Bilbao
  - Hospital Parc Taulí, Sabadell

IPD SHARING:
Plan to Share IPD: No